CLINICAL TRIAL: NCT05114174
Title: Evaluation and Implementation of an mHealth Intervention to Prevent Gestational Obesity in the Metropolitan Region and the Aconcagua Valley.
Brief Title: Evaluation and Implementation of an mHealth Intervention Called Mami-educ to Fight Against Gestational Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Sebastián (Other)
Collaborators: Universidad de Valparaiso (Other); Fondo de Fomento al Desarrollo Científico y Tecnológico, Fondef. (Unknown)
Responsible Party: Principal Investigator, Delia Indira Chiarello, Investigator Ph.D., Universidad San Sebastián
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SA21I0099
Record Dates: First submitted 2021-10-15; First posted 2021-11-09 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2022-10

CONDITIONS: Gestational Weight Gain; Obesity, Maternal
Keywords: mHealth; Gestational obesity; Social theory
MeSH Terms: conditions — Gestational Weight Gain; Pregnancy in Obesity

STUDY DESIGN:
Intervention Model Description: Classic randomized clinical trial (RCT).
Who Masked: Care Provider
Masking Description: Blinding will be done in a single-blind fashion. The care provider will be blinded to the randomization of the subjects to avoid bias in routine care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care group (No Intervention): Pregnant women enrolled in the prenatal control program who receive routine medical care.
- mami-educ group (Experimental): Pregnant women enrolled in the prenatal care program who receive routine medical care and nutritional messages mom-educ.
  Interventions: Other: mami-educ

INTERVENTIONS:
Other: mami-educ — The intervention corresponds to sending 3 messages a week through Telegram, with nutritional information, for 12 consecutive weeks (a different nutritional topic each week). The messages address the three domains of learning, cognitive, affective, and psychomotor for each topic.
  Arms: mami-educ group

SUMMARY:
The World Federation of Obesity warns that the main health problem of the next decade will be childhood obesity. Furthermore, obesity and its consequences have been reported to originate in intrauterine life. Gestational obesity produces profound effects on fetal genome programming, thereby inducing changes in prenatal metabolism that extend to the postnatal period, which is also associated with increased susceptibility to developing cardiovascular and metabolic diseases in adulthood.

Excessive maternal weight gain early in pregnancy has been repeatedly associated with increased adiposity in childhood and adolescence of its offspring. Obesity is a complex phenomenon influenced by social determinants of health, which include demographic, socioeconomic, behavioral, environmental, and genetic factors. At the primary prevention level, nutrition constitutes a modifiable risk factor during pregnancy. Therefore establishing healthy nutritional behaviors during the first trimester of pregnancy is key to the primary prevention of the intergenerational transmission of obesity.

New ways of approaching the target population are required to maintain nutritional recommendations as a priority in the daily decision-making (top of mind) of pregnant women. For many women, this period is a powerful motivator for self-care.

Interventions based on behavioral theories provide a better understanding of the underlying mechanisms that determine health-related behavior change and have the potential to be more effective in promoting adherence to weight gain control. Social Cognitive Theory (TCS) is an integrated model of behavior change commonly applied in mobile health interventions that address diet, physical activity or weight loss.

Mobile health programs (mHealth) are potentially more effective than face-to-face interventions, especially during a public health emergency like the COVID-19 outbreak. This proposal intends to "deliver" messages with evidence-based information directly to pregnant women, in order to influence their nutritional behavior to avoid excessive gestational weight gain.

The hypothesis of this proposal is that the mHealth intervention called "mami-educ", which consists of sending messages with nutrition counseling during pregnancy through the Telegram platform, is effective in reducing excessive gestational weight gain in pregnant women attending Family Health Care Centers in an urban and predominantly rural area.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who receive care in the 6 CESFAMs of El Bosque and Aconcagua Valley over 18 years of age; pregnant women with gestational age ≤ 12 weeks of gestation (first trimester)
* Pregnant women with a single pregnancy
* Healthy pregnant women
* Chilean or immigrant women who speak Spanish
* The participants must have a mobile device that allows the use of the Telegram application
* Pregnant women who agree to be randomized
* Pregnant women who have voluntarily signed the informed consent to participate in this study

Exclusion Criteria:

* A multiple pregnancy
* Conditions that require a special diet
* Participants with psychiatric illness or other pre-pregnancy pathology
* History of recurrent abortions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain | Nine months
  Maternal weight gain measure in kilograms by month

SECONDARY OUTCOMES:
Maternal outcome | Nine months
  Medical diagnosis of of either preeclampsia, gestational diabetes or gestational hypertension
Perinatal outcome | At birth
  Labor delivery week
Apgar score | At birth
  Apgar score report
Newborn birth weight | At birth
  Newborn birth weight measure in grams

CONTACTS AND LOCATIONS:
Overall Officials: Delia I Chiarello, Ph.D, Study Director — Universidad San Sebastián
Locations (2):
- Chile (2):
  - Delia I Chiarello, Santiago, Providencia
  - Fabián Pardo, San Felipe, Región de Valparaíso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiarello DI, Pardo F, Moya J, Pino M, Rodriguez A, Araneda ME, Bertini A, Gutierrez J. An mHealth Intervention to Reduce Gestational Obesity (mami-educ): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Feb 15;12:e44456. doi: 10.2196/44456. PMID 36790846